CLINICAL TRIAL: NCT03059186
Title: A Randomised Controlled Trial of a Brief Gratitude Intervention in Improving Well-being and Coping in People Living With Inflammatory Bowel Disease
Brief Title: A Gratitude Intervention in Improving Well-being and Coping in People Living With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Peter Isebor, Principal Investigator, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 151209
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Online daily gratitude journal.
  Interventions: Behavioral: Gratitude diary
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Gratitude diary — The intervention involves keeping a record of three things that the individual feels grateful for during that day.
  This can be completed daily, and for the purpose of this study will be completed every evening for the duration of one week.
  Other Names: Count your blessings
  Arms: Intervention

SUMMARY:
The primary aim of the proposed research is to investigate the extent to which a one-week online gratitude intervention can improve levels of wellbeing in individuals living with Inflammatory Bowel Disease (IBD). A secondary aim was to investigate the extent to which dispositional gratitude influences levels of coping and wellbeing and to what extent this mediates the effect of the intervention. Participants with IBD will be randomized to either treatment or control group. Participants will complete measures pre- and post- intervention, and follow-up (eight weeks) measuring: gratitude (state and trait), illness severity, mood, stress and coping.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of inflammatory bowel disease from a clinician.

Exclusion Criteria:

* No access to internet via smartphone, tablet or computer.
* Cannot read English

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change in The Depression Anxiety and Stress Scale- 21 | 1 week, and 8 weeks follow up.
  Change in wellbeing
Change in the Inflammatory Bowel Disease Questionnaire UK | 1 week, and 8 weeks follow up
  Change in health

SECONDARY OUTCOMES:
Change in the IBD Self-efficacy scale | 1 week and 8 weeks follow up
  Change in coping
Change in the Gratitude Questionnaire 6 | 1 week and 8 weeks follow up
  Change in gratitude
Change in the Gratitude Adjectives Checklist | 1 week and 8 weeks follow up
  Change in gratitude
Change in Emotion Regulation Questionnaire-Revised | 1 week and 8 weeks
  Change in emotion regulation

CONTACTS AND LOCATIONS:
Overall Officials: Georgina Rowse, Dr, Study Chair — Researcher/Supervisor; Amrit Sinha, Study Chair — Research Support Secretary
Locations (1):
- University of Sheffield Clinical Psychology Department Catherdral Court, Sheffield, United Kingdom

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391